CLINICAL TRIAL: NCT06691321
Title: Efficacy of Caspofungin for Pneumocystis Jirovecii Pneumonia in People Living With HIV/AIDS.
Brief Title: Caspofungin for Pneumocystis Pneumonia in PLWHIV.
Status: Recruiting | Type: Observational
Sponsor: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Principal Investigator, Santiago Avila-Rios, Head of the Center for Research in Infectious Diseases., Instituto Nacional de Enfermedades Respiratorias
Other Study IDs: C35-23
Record Dates: First submitted 2024-11-11; First posted 2024-11-15 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: HIV-1-infection; Pneumocystis Pneumonia
Keywords: Pneumocystis jirovecii pneumonia; Echinocandins; Caspofungin
MeSH Terms: conditions — Pneumonia, Pneumocystis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TMP/SMZ (Control): Patients with HIV and PCP starting treatment with trimethoprim/sulfamethoxazole (TMP/SMZ).
- Caspo (Study): Patients with HIV and PCP starting treatment with caspofungin with or without clindamycin or primaquine; or switching from trimethoprim/sulfamethoxazole to caspofungin before day 7 of treatment initiation.

SUMMARY:
Pneumocystis jirovecii pneumonia is a significant concern in peaple with HIV/AIDS, often severe and potentially fatal. While trimethoprim/sulfamethoxazole remains the primary treatment, safety concerns exist with alternative options. Research on Pneumocystis jirovecii's beta-D glucan composition has prompted investigations into echinocandins like caspofungin, showing promise in murine models and some positive results in human studies. Evaluating caspofungin's efficacy through observational studies is crucial due to safety advantages over current treatments and limited documented data.

DETAILED DESCRIPTION:
Pneumocystis jirovecii pneumonia (PCP) is a significant opportunistic disease in immunocompromised patients with HIV/AIDS, becoming increasingly prevalent. This condition can range in severity, at times being fatal and necessitating drastic measures. The standard first-line treatment, trimethoprim/sulfamethoxazole, has been unchanged for over three decades. While other drugs have been approved as second-line treatments, they come with safety concerns such as increased risk of hypersensitivity reactions and adverse effects.

Research on Pneumocystis jirovecii has faced challenges due to difficulties in cultivation, requiring in vivo models for study. Previous studies have found that the wall of Pneumocystis spp. contains beta-D glucans in one phase of its life cycle. This discovery has led to investigations into the effectiveness of echinocandins, specifically caspofungin, on Pneumocystis spp. Promising results have been observed in murine models; however, these studies were conducted on species that do not affect humans. Clinical observational studies in humans have shown positive response and safety, albeit using caspofungin in combination with other drugs rather than as monotherapy.

Considering the superior safety profile of echinocandins compared to first-line treatments for P. jirovecii, and the limited documented data in case reports or series, it is important to assess the efficacy of caspofungin in observational studies to address this gap.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable or proven PCP, according to its diagnostic classification (refer to classification at the end of this section).
* Have clinical laboratory and virological diagnostic laboratory studies at the time of admission.

  * Classification criteria for Pneumonia by P. jirovecii according to Robert-Gangneux et al.:

Proven: Confirmation by pathology or microbiology. Possible: Presence of three out of four clinical or radiological criteria. Probable: Presence of one clinical or radiological criterion without another identified microorganism.

Exclusion Criteria:

* With a treatment switch to caspofungin after day 7 of treatment initiation (applies only to group B).
* Patients who have developed an additional opportunistic lung infection during their hospitalization, other than cytomegalovirus pneumonitis or SARS-CoV-2 pneumonia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will be conducted with data extracted from the clinical records of patients with human immunodeficiency virus (HIV), hospitalized for Pneumocystis jirovecii pneumonia (PCP) from January 2015 to December 2023.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Mortality by group at a 30-day follow up. | 30 days
  Compare the efficacy of caspofungin-based treatment with trimethoprim/sulfamethoxazole on 30-day mortality in hospitalized patients with Pneumocystis jirovecii pneumonia.

SECONDARY OUTCOMES:
Mortality by group at a 90-day follow up. | 90 days
  Compare the efficacy of caspofungin-based treatment with trimethoprim/sulfamethoxazole on 90-day mortality in hospitalized patients with Pneumocystis jirovecii pneumonia.
Length of hospital stay per group. Length of hospital stay per group. Length of hospital stay per group. Length of hospital stay per group. | 90 days
  Compare the length of hospital stay between the groups.
Requirement and duration of high-flow nasal cannula. Requirement and duration of high-flow nasal cannula between groups. | 90 days
  Compare the requirement and duration of high-flow nasal cannula between the groups.
Requirement and duration of invasive mechanical ventilation. | 90 days
  Compare the requirement and duration of invasive mechanical ventilation between the groups.
Acute respiratory distress syndrome incidence. | 90 days
  Compare the incidence of acute respiratory distress syndrome during hospitalization.
Adverse events. | 90 days
  Determine the incidence of adverse reactions to the different regimens used as treatment for PCP.

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Avila, PhD, Principal Investigator — Center for Research in Infectious Diseases (CIENI)
Locations (1):
- Center for Research in Infectious Diseases (CIENI), Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: Yes
It is planned to publish the database used for the statistical analysis, including only the variables utilized for the manuscript(s) submitted for publication. These databases will be shared according to the specifications of the journal to which they have been submitted.
Supporting Information: SAP, Analytic Code
Time Frame: These databases will be shared once the manuscript(s) have been accepted for publication in a journal and will remain open indefinitely.
Access Criteria: The databases will be available in a public repository or as a downloadable file attached to the publication.

REFERENCES:
- [Background] Robert-Gangneux F, Belaz S, Revest M, Tattevin P, Jouneau S, Decaux O, Chevrier S, Le Tulzo Y, Gangneux JP. Diagnosis of Pneumocystis jirovecii pneumonia in immunocompromised patients by real-time PCR: a 4-year prospective study. J Clin Microbiol. 2014 Sep;52(9):3370-6. doi: 10.1128/JCM.01480-14. Epub 2014 Jul 9. PMID 25009050
- [Background] Tian Q, Si J, Jiang F, Xu R, Wei B, Huang B, Li Q, Jiang Z, Zhao T. Caspofungin combined with TMP/SMZ as a first-line therapy for moderate-to-severe PCP in patients with human immunodeficiency virus infection. HIV Med. 2021 Apr;22(4):307-313. doi: 10.1111/hiv.13013. Epub 2020 Dec 4. PMID 33277811
- [Background] Huang Y, He X, Chen H, Harypursat V, Lu Y, Yuan J, Nie J, Liu M, Yu J, Zhang Y, Jiang Z, Qin Y, Xu L, Zhou G, Zhang D, Chen X, Zheng B, Chen Y. No Statistically Apparent Difference in Antifungal Effectiveness Observed Among Trimethoprim/Sulfamethoxazole Plus Clindamycin or Caspofungin, and Trimethoprim/Sulfamethoxazole Monotherapy in HIV-Infected Patients with Moderate to Severe Pneumocystis Pneumonia: Results of an Observational Multicenter Cohort Study. Infect Dis Ther. 2022 Feb;11(1):543-557. doi: 10.1007/s40121-021-00586-5. Epub 2022 Jan 20. PMID 35050490
- [Background] Cushion MT, Linke MJ, Ashbaugh A, Sesterhenn T, Collins MS, Lynch K, Brubaker R, Walzer PD. Echinocandin treatment of pneumocystis pneumonia in rodent models depletes cysts leaving trophic burdens that cannot transmit the infection. PLoS One. 2010 Jan 29;5(1):e8524. doi: 10.1371/journal.pone.0008524. PMID 20126455
- [Background] Armstrong-James D, Stebbing J, John L, Murungi A, Bower M, Gazzard B, Nelson M. A trial of caspofungin salvage treatment in PCP pneumonia. Thorax. 2011 Jun;66(6):537-8. doi: 10.1136/thx.2010.135350. Epub 2010 Sep 29. No abstract available. PMID 20880871
- [Background] Walzer PD, Schultz MG, Western KA, Robbins JB. Pneumocystis carinii pneumonia and primary immune deficiency diseases of infancy and childhood. J Pediatr. 1973 Mar;82(3):416-22. doi: 10.1016/s0022-3476(73)80114-3. No abstract available. PMID 4540607
- [Background] Lobo ML, Esteves F, de Sousa B, Cardoso F, Cushion MT, Antunes F, Matos O. Therapeutic potential of caspofungin combined with trimethoprim-sulfamethoxazole for pneumocystis pneumonia: a pilot study in mice. PLoS One. 2013 Aug 5;8(8):e70619. doi: 10.1371/journal.pone.0070619. Print 2013. PMID 23940606
- [Background] Sun P, Tong Z. Efficacy of caspofungin, a 1,3-beta-D-glucan synthase inhibitor, on Pneumocystis carinii pneumonia in rats. Med Mycol. 2014 Nov;52(8):798-803. doi: 10.1093/mmy/myu060. Epub 2014 Oct 6. PMID 25288652
- [Background] Skalski JH, Kottom TJ, Limper AH. Pathobiology of Pneumocystis pneumonia: life cycle, cell wall and cell signal transduction. FEMS Yeast Res. 2015 Sep;15(6):fov046. doi: 10.1093/femsyr/fov046. Epub 2015 Jun 12. PMID 26071598